CLINICAL TRIAL: NCT02392195
Title: Brain Characteristics Noted Prior to and Following Treatment of Deformational Plagiocephaly With a Helmet
Brief Title: Brain Characteristics Noted Prior to and Following Treatment
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michele DeGrazia, Director Nursing Research NICU, Boston Children's Hospital
Other Study IDs: IRB-P00004233
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Nonsynostotic Plagiocephaly
Keywords: Plagiocephaly
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Plagiocephaly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single arm; Non-interventional: A convenience sample of 10-15 infants born at term gestation, that are </= 6 months of age with significant DP (defined as head flattening requiring helmet therapy) and no major health issues will be recruited into this phase 1 descriptive pilot study
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Observational

SUMMARY:
This study will enable investigators to find out if brain structure and characteristics are affected by the shape of the infant's head, and if changes in the brain occur with helmet therapy.

DETAILED DESCRIPTION:
A dramatic increase in the number of infants diagnosed with Deformational Plagiocephaly (DP) has been observed worldwide since institution of the American Academy of Pediatrics' Back to Sleep Program. According to one published report, the incidence of DP ranges between 3-48%; this translates into120,000-2 million infants/year who develop DP in the United States alone. Some healthcare providers believe that DP is a purely cosmetic condition. This mindset undermines the importance of prevention and correction. In New Zealand, a recent study demonstrated that 39% of children without corrective action had persistent DP at age 3 to 4 years. Additionally, several studies have demonstrated associations between impaired social interactions, developmental problems and DP.Thus some researchers now believe that there may be a spectrum of untoward outcomes from brain remodeling resulting from DP. Recent technological advances now allow the detection of diminutive changes in brain structure. In this multidisciplinary descriptive pilot study we will use brain MRI (Magnetic Resonance Imaging) and a cerebral tissue oxygenation monitor, namely Frequency Domain Near Infrared and Diffuse Correlation Spectroscopy (FDNIR/DCS) to describe if differences in brain structure and characteristics exist in infants with significant DP before and after correction of the deformational defect. This study will enable investigators to seek preliminary evidence that brain development is influenced by the shape of the cranial vault, and that changes in brain structure and characteristics occur with helmet therapy. Additionally this study will help to determine the need for a larger investigation of this phenomenon that would further establish an association between DP and developmental delay.

ELIGIBILITY:
Inclusion Criteria:

1. - DP requiring helmet therapy
2. -Term gestation at birth (37 weeks or greater)
3. -Less than/or equal to 8 months of age
4. -No history of major health problem such as birth injury, genetic disorder, intracranial hemorrhage, hydrocephalus, neurologic abnormality
5. -No history of implantable metal device or internal/external orthotic device

Exclusion Criteria:

1. - DP not requiring helmet therapy
2. -Premature gestation at birth (less than 37 weeks gestation).
3. -Greater than 8 months of age
4. -History of major health problem such as birth injury genetic disorder, intracranial hemorrhage, hydrocephalus, neurologic abnormality
5. -History of implantable metal device or internal/external orthotic device
6. -Infants not completing prescribed treatment for correction with a helmet

Max Age: 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Deformational Plagiocephaly in full term, healthy infants.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele DeGrazia, PhD, RN, NNP, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm; Non-interventional
Started | 10
Completed | 2
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Single Arm; Non-interventional: A convenience sample of infants born at term gestation, </= 6 months of age with significant Deformational Plagiocephaly (DP) (defined as head flattening requiring helmet therapy) and no major health issues will be recruited into this phase 1 descriptive pilot study
  Non-interventional: Observational
Arm/Group | Single Arm; Non-interventional
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: months] | 6 [5 to 7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Cranial vault asymmetry index (CVAI) > 8.75% [Count of Participants; unit: Participants] — Cranial vault asymmetry (CVA): the absolute difference in cranial diagonals.
  Cranial vault asymmetry (CVAI): measure of cranial vault asymmetry in relationship to the overall size of the head, it is the difference between the diagonals divided by the longer of the diagonals multiplied by 100.
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Qualitatively Determined Normalization of White Matter Pathways
Description: We will compare if nerve pathways are appreciably different in the area of head flattening following helmet therapy by visual examination and comparison of areas of asymmetry vs. symmetry.
Time Frame: 2-6 months
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm; Non-interventional: A convenience sample of infants born at term gestation, that are </= 6 months of age with significant DP (defined as head flattening requiring helmet therapy) and no major health issues will be recruited into this phase 1 descriptive pilot study
  Non-interventional: Observational
Arm/Group | Single Arm; Non-interventional
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Number of Participants With Improved Developmental Exams Post Helmet Therapy
Description: The Mullen (Scales of Early Learning) was used to determine developmental scores. This tool provides a profile of cognitive ability in five areas:
  Gross Motor, Fine Motor, Expressive Language, Receptive Language, and Visual Reception. Each of the 5 assessment that has a raw score that is then given a percentile rank and descriptive category (below average, average, above average) for interpretation purposes. Descriptive categories pre treatment were compared to post treatment to determine if scores had improved.
Time Frame: 2-6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm; Non-interventional
Number analyzed (Participants) | 2
Participants | 2

3. Other Pre Specified Outcome: Number of Participants With Improved Cranial Asymmetry After Cranial Orthotic Treatment
Description: Cranial asymmetry was assessed using the Cranial Vault Asymmetry Index (CVAI). MRI's were utilized to determine CVAI. Asymmetry pre treatment was compared to post treatment to see if asymmetry improved.
Time Frame: Collected retrospectively
Measure: Number; unit: participants
Arm/Group | Single Arm; Non-interventional
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Arm; Non-interventional
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT02392195/Prot_SAP_000.pdf